CLINICAL TRIAL: NCT05821478
Title: A Multicentric Randomized Double-Blind Phase 3 Trial Evaluating the Efficacy of an Adapted Antibiotherapy in Hurley Stage 2 Active Hidradenitis Suppurativa Patients Versus Tetracycline Derivative
Brief Title: Efficacy of an Adapted Antibiotherapy in Hurley Stage 2 Hidradenitis Suppurativa Patients
Acronym: ABCESS2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Centre Hospitalier Universitaire de Caen (Other); Hôpital Necker-Enfants Malades (Other); Ministry of Health, France (Other Government); Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-018
Record Dates: First submitted 2019-04-16; First posted 2023-04-20 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Antibioresistance; Antibiotherapy
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Ceftriaxone; Metronidazole; Rifampin; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Multicentric randomized double-blind phase 3 trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental treatment (Experimental): a 3-week course of ceftriaxone (Rocephin) IV injection (daily dose 2g/day)
  + oral metronidazole (daily dose 1500mg) followed by a 3-week course of oral rifampicin (Rifadin with 10mg/kg/day) + moxifloxacin (Izilox daily dose 400mg) + metronidazole (daily dose 1500mg) followed by a 6-week course of oral rifampicin (Rifadin with 10mg/kg/day) + moxifloxacin (Izilox daily dose 400mg).
  A placebo for lymecycline will also be administered during this intensive treatment phase
  Interventions: Drug: ROCEPHIN, metronidazole, RIFADIN, IZILOX, placebo combination therapy
- Control (Active Comparator): 12-week course of oral lymecycline (Tetralysal daily dose 452mg) Placebos for all experimental drugs will also be administered during this intensive treatment phase
  Interventions: Drug: Lymecyclin and corresponding placebos of the experimental arm

INTERVENTIONS:
Drug: ROCEPHIN, metronidazole, RIFADIN, IZILOX, placebo combination therapy — a 3-week course of ceftriaxone injection + oral metronidazole followed by a 3-week course of oral rifampicin + moxifloxacin +metronidazole followed by a 6-week course of oral rifampicin + moxifloxacin
  Other Names: Experimental treatment
  Arms: Experimental treatment
Drug: Lymecyclin and corresponding placebos of the experimental arm — 12-week course of oral lymecycline.
  Other Names: Control treatment
  Arms: Control

SUMMARY:
The study evaluates the efficacy of an adapted antibiotherapy in Hurley stage 2 active Hidradenitis Suppurativa patients versus tetracycline derivative

DETAILED DESCRIPTION:
The antibiotic strategy is targeted against specific pathobionts which have been identified in HS lesions by the investigator's team.

Half of participants will receive a 3-week course of ceftriaxone + metronidazole treatment followed by 3 weeks of rifampicin + moxifloxacin + metronidazole combination, then 6 weeks of rifampin + moxifloxacin (experimental groupe), versus a 12 weeks course of lymecycline (control group) Double blind treatment phase will stop at week 12. All patients whatever their randomization arm or their remission status will begin follow-up treatment according to standard care recommendations (Société Française de Dermatologie): lymecycline, doxycycline or cotrimoxazole. Prescription will be upon decision of the investigator.

This maintenance treatment is not experimental.

ELIGIBILITY:
Inclusion Criteria:

* Adults < 60 years old
* Diagnosis of HS according to European Dermatology guidelines:

  * Recurrent inflammation occurring more than 2 times in the past 6 months in the inverse regions of the body, presenting with nodules, sinus-tracts and/or scarring.
  * Signs: Involvement of axilla, genitofemoral area, perineum, gluteal area (and infra-mammary areafor women). Presence of nodules (inflamed or noninflamed), sinus tracts (inflamed or noninflamed), abscesses, scarring (atrophic, mesh-like, red, hypertrophic or linear)
* Active HS with i) ≥ 1 year of evolution and ii) ≥ 4 flares during the previous year
* Clinical severity of HS at inclusion: Hurley stage 2
* BMI < 35
* Written informed consent from patient
* Patient able to complete DLQI
* Patients affiliated to the French health system (Assurance Maladie), except French state medical aid beneficiaries (Aide Médicale d'Etat)
* Active compatible contraception for men and women of childbearing or inability to procreate
* Available laboratory blood test performed within the last 2-months

Non inclusion Criteria:

* Person < 18 and ≥ 60 years old
* Former stage 3 HS
* Previous use of the experimental treatment
* Unauthorized drugs for the study during the month preceding the inclusion
* Any contra-indication to study treatments or excipient (e.g. lactose, cornstarch, riboflavin notably):

pregnancy, breastfeeding, known allergy to experimental or reference drugs, wheat allergy, tendinopathy, QT prolongation, bradycardia, heart failure, heart rhythm disturbances, hydroelectrolytic disorders, hypokalemia, coagulation disorders, severe liver/kidney dysfunction, porphyria, mandatory use of nonsteroidal anti-inflammatory drugs (NSAIDs) for other medical conditions

* Unbalanced diabetes (ie HbA1c above 7%)
* Dysphagia, untreated gastro-oesophageal reflux/ulcer
* BMI ≥ 35
* Immune suppression, inflammatory disease, including gastroenterologic and rheumatologic inflammatory conditions
* Lactase deficiency, lactose and galactose intolerance
* Malabsorption syndrome
* Person living in the same household as another patient
* Person under guardianship or curatorship
* Individuals with any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives (e.g patient unable to complete DLQI, or poor predictable observance
* Participation in another interventional research on health products studies
* Patients requiring repeated (more than 3/year) use of antibiotics for a chronic disease other than HS
* Alcohol-dependant patients defined as an addiction to alcohol with a negative impact on health, social or personal life

Exclusion criteria:

Pregnancy QT prolongation Abnormal result of routine lab tests corresponding to contra-indication to study treatments Unauthorized drug for the study during all the study (from study treatments interactions listed in the SmPC, Cf. unauthorized drug listed in non-inclusion criteria).

Development of hypersensitivity to any of the study products and/or excipients (e.g. lactose, corn starch, riboflavin).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-27 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients reaching clinical remission at week 12, defined by an improvement of 90% of the IHS4 score from the baseline (IHS4 (1)) | at week 12
  The clinical remission is defined as a 90% improvement of the International Hidradenitis Suppurativa Severity Score (IHS4) at week 12 compared to the baseline.
  The IHS4 score is a validated composite score developped to assess dynamically HS severity (1). It is calculated by adding the number of inflammatory nodules to the number of abscesses multiplied by 2 and to the number of draining tunnels multiplied by 4. A total score of 3 or less corresponds to mild severity HS, 4-10 to moderate severity HS and 11 or higher to severe disease.

SECONDARY OUTCOMES:
Change in Physician Global Assessment (PGA) | from baseline to week 52
  Physician assessment describe by differents severity : from Clear (no nodule) to Very severe (more than 5 abscesses or fistulas) Score evaluated at baseline / week 6 / week 12/ week 24/ week 52
Change in Modified Sartorius score | from baseline to week 52
  Score calculated by points from 0 (better) with differents parameters involved such as location / number / size / type of lesions Score evaluated at baseline / week 6 / week 12/ week 24/ week 52
Change in Hurley Score | from baseline to week 52
  Score described with 3 stages from I (less severity) to III (most severe) Score evaluated at baseline / week 6 / week 12/ week 24/ week 52
Change in Hidradenitis Suppurativa Severity Score (IHS4) score | from baseline to week 52
  Score calculated by points from <3pts (Mild) to > 11pts (Severe) by nb of nodules, nb of abscesses and nb of draining tunnels Score evaluated at baseline / week 6 / week 12/ week 24/ week 52
Change in Hidradenitis Suppurativa Clinical Response (HiSCR) score | from baseline to week 52
  Global Assessment score of clear, minimal, or mild evaluated by (i) at least a 50% reduction in AN (abscess and nodule count), (ii) no increase in the number of abscesses and (iii) no increase in the number of draining fistulas from baseline Score evaluated at baseline / week 6 / week 12/ week 24/ week 52
Change in Dermatology Life Quality Index (DLQI) score (Patient's HS evaluation) | from baseline to week 52
  Evaluated with the Dermatology Life Quality Index (DLQI) Score calculated by points from 0 to 30 following patient answers on quality of life questions Score evaluated at baseline / week 6 / week 12/ week 24/ week 52
Change of patient pain | from baseline to week 52
  Intensity of pain evaluated with the visual analog scale (VAS) from 0 (no pain) to 10 (pain as bad as it could possible be) Score evaluated at baseline / week 6 / week 12/ week 24/ week 52
Microbiological bacterial Change on the worst lesion microbiome at W12 | at baseline and week 12
  By identification of microbiology bacterial metagenomics (by skin lesional swab sample)
Microbiological metagenomics Change on the worst lesion microbiome at W12 | at baseline and week 12
  By identification of multidrug resistant bacteria (by rectal swab sample)
Number of pain killers received by patients | from baseline to week 52
  Number of pain killers prescribed for flares (acute worsening of one or more HS lesions)
Number of antibiotic treatments received by patients | from baseline to week 52
  Number of antibiotic treatments prescribed for flares (acute worsening of one or more HS lesions)
Time without flare of HS | from baseline to week 52
  Evaluated by number of flares reported or not using a patient journal
Change in BMI | from baseline to week 52
  Calculated by combined weight and height measures
Abnormal biological value of Hemoglobin | from baseline to week 12
  measured in g/L, compared to normal ranges
Abnormal biological value of white cells | from baseline to week 12
  measured in units of cells / mm3 , compared to normal ranges
Abnormal biological value of neutrophils | from baseline to week 12
  measured in units of cells / mm3 , compared to normal ranges
Abnormal biological value of platelet count | from baseline to week 12
  measured in units of cells / mm3 , compared to normal ranges
Abnormal value of AST liver enzyme | from baseline to week 12
  AST value > 4 x Upper limit of normal
Abnormal value of ALT liver enzyme | from baseline to week 12
  ALT value > 4 x Upper limit of normal
Number of adverse events of all kind | from baseline to week 52
  AE defined by SOC and PT according to MedDra dictonnary
Non complete drug administration | from baseline to week 12
  Evaluated by total number of capsules not taken according to patient journal

CONTACTS AND LOCATIONS:
Overall Officials: Maïa Delage-Toriel, MD, Principal Investigator — Institut Pasteur
Locations (4):
- France (4):
  - Hôpital de la Timone, Marseille
  - Centre Médical de l'Institut Pasteur, Paris
  - Hopital St Joseph, Paris
  - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: CSR
Time Frame: After publication, for 25 years
Access Criteria: By publication in scientific journals and / or presented in scientific or medical meetings

REFERENCES:
- [Background] Guet-Revillet H, Jais JP, Ungeheuer MN, Coignard-Biehler H, Duchatelet S, Delage M, Lam T, Hovnanian A, Lortholary O, Nassif X, Nassif A, Join-Lambert O. The Microbiological Landscape of Anaerobic Infections in Hidradenitis Suppurativa: A Prospective Metagenomic Study. Clin Infect Dis. 2017 Jul 15;65(2):282-291. doi: 10.1093/cid/cix285. PMID 28379372
- [Background] Guet-Revillet H, Coignard-Biehler H, Jais JP, Quesne G, Frapy E, Poiree S, Le Guern AS, Le Fleche-Mateos A, Hovnanian A, Consigny PH, Lortholary O, Nassif X, Nassif A, Join-Lambert O. Bacterial pathogens associated with hidradenitis suppurativa, France. Emerg Infect Dis. 2014 Dec;20(12):1990-8. doi: 10.3201/eid2012.140064. PMID 25418454
- [Background] Join-Lambert O, Coignard H, Jais JP, Guet-Revillet H, Poiree S, Fraitag S, Jullien V, Ribadeau-Dumas F, Theze J, Le Guern AS, Behillil S, Lefleche A, Berche P, Consigny PH, Lortholary O, Nassif X, Nassif A. Efficacy of rifampin-moxifloxacin-metronidazole combination therapy in hidradenitis suppurativa. Dermatology. 2011 Feb;222(1):49-58. doi: 10.1159/000321716. Epub 2010 Nov 25. PMID 21109728